CLINICAL TRIAL: NCT03900689
Title: Defining Personal and Communal Aspects of Social Determinants of Health in Glioblastoma Population
Brief Title: Social Determinants of Health in Glioblastoma Population
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00057185; WFBCCC 03119 (Other: Wake Forest Baptist Comprehensive Cancer Center); NCI-2019-02214 (Other: Clinical Trials Reporting Program)
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Glioma; Astrocytoma; Oligodendroglioma; Ependymoma; Ganglioglioma; Pleomorphic Xanthoastrocytoma
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma; Ependymoma; Ganglioglioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health Services Research - Part 1 Survey: Participants will be asked to complete a series of surveys. This will be preferentially completed on the same day of the visit but may be completed at a subsequent visit, over the telephone or taken home and sent back to the clinic.
  Interventions: Other: Part 1 Survey Group
- Health Services Research - Part 2 - Focus Group: Patients identified in Part 1 will be offered participation in the focus groups in Part 2. All patients enrolled in Part 1 will be considered for participation in Part 2. Approximately 30 total patients will be invited to participate. Patients who agree to be contacted will receive a telephone call or contacted in clinic and invited to participate in the Part 2 focus group.
  Interventions: Other: Part 2 Focus Group

INTERVENTIONS:
Other: Part 1 Survey Group — At the first study visit, participants will answer a series of survey questions about their neighborhoods, educational levels, social activities, access to transportation and food, healthcare management and where participants find social and spiritual support. General information such as age, ethnicity and address will also be collected.
  Groups: Health Services Research - Part 1 Survey
Other: Part 2 Focus Group — If participants from Part 1 agree to be contacted for Part 2, participants will be included in a focus group to explore unexpected findings and further investigate social determinants identified in Part 1.
  Groups: Health Services Research - Part 2 - Focus Group

SUMMARY:
The overall aim of this study is to prospectively characterize social health disparities in a cross-sectional cohort of glioma patients with attention to exploring and thematically categorizing the patient-specific and community-level factors. This will be conducted in two parts.

DETAILED DESCRIPTION:
Part 1:

Primary Objectives

1. To describe the social determinants of health in a cross-section of patients with WHO Grade 2-4 gliomas using a group of validated instruments including the PRAPARE instrument, the Accountable Health Communities Health-Related Social Needs Screening Tool (AHC HRSN), and supplementary questions.

Secondary Objectives

1. To compare social determinants of health between patients residing in economically disadvantaged and advantaged communities as defined in our prior study (low income communities vs high income county communities, by zip code).
2. To compare social determinants of health between patients residing in economically disadvantaged and advantaged communities as defined by other means including county (low income communities vs high income communities, by county), by urban vs rural (urban vs rural, by city), and by area deprivation index (see Section 5.2).
3. To quantify and compare the patient- and community-level social determinants of health present in the cohort and by community (low income community vs high income community).
4. To compare the time to presentation, time to treatment initiation, and extent of surgery for patients from economically disadvantaged and advantaged communities as described above.

Part 2:

Data from our preliminary study revealed differences in survival for patients from low income communities compared to high income community zip codes. The overarching goal of Part 2 is to further characterize the social factors that characterize low income community and high income communities and may contribute to the differences in outcome.

Primary Aim

1. To identify, compare, contrast, and contextualize the patient- and community-specific social determinants for patients residing in (1) low income communities and high income community zip codes and (2) urban and rural communities.
2. To explore how patients perceive communication with their providers about social and community factors that contribute to health outcomes and understand the barriers, challenges, and opportunities to improve patient-provider communication.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Adults who are 18 years or older
* Have a histologically confirmed glioma of any grade (WHO Grade 2-4: astrocytoma, oligodendroglioma, ependymoma, ganglioglioma, pleomorphic xanthroastrocytoma)
* Currently receiving primary oncologic care at Wake Forest Baptist Comprehensive Cancer Center
* Have the ability to speak and read either English or Spanish.
* Ability to provide informed consent

Part 2:

* Participants who participated in Part 1 and express willingness to be contacted about Part 2
* Ability to provide informed consent
* Ability to speak and understand English

Inclusion of Women and Minorities (for Part 1 and Part 2)

• Women of all races and ethnicity who meet the above-described eligibility criteria are eligible for this trial.

Exclusion Criteria:

• Patients who are unable to read or complete the required study-related forms. Patients who are unable to read but can be assisted by a proxy or family member will be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a two part, sequential, mixed-methods study. Part 1 will enroll a cross-section of glioma patients at Wake Forest Baptist Comprehensive Cancer Center. In part 2, participants from Part 1 will be identified, selected, and invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2022-03-27 (Actual)

PRIMARY OUTCOMES:
PRAPARE Instrument Questionnaire | Approximately 30 minutes
  A 21 question questionnaire to collect data based on five main social determinants of health (education, economic status, neighborhood/surrounding environment, health and healthcare, community involvement). The questionnaire is comprised of Yes or No answers, multiple choice questions and Likert scale questions (not at all to quite a bit). This will be completed in Part 1 of the study.
Accountable Health Communities Health-Related Social Needs Screening Tool | Approximately 30 minutes
  An 18 question screening tool to help find out participants' needs in areas of housing instability, food insecurity, utility help needs, financial status, family and community support and physical activity. The questionnaire is comprised of Yes or No answers, multiple choice questions and Likert scale questions (Not hard at all to very hard; never to often). This will be completed in Part 1 of the study.
Social Determinants of Health Supplementary Questionnaire | Approximately 30 minutes
  The questionnaire is composed of 5 sections (economic status, social and community context, neighborhood and environment, health and healthcare and education) and has a combination of Yes or No questions, multiple choice questions, and Likert questions (never to always). This will be completed in Part 1 of the study.

SECONDARY OUTCOMES:
Proportion of Social Determinants Based on Two Communities | Approximately 90 minutes
  Social determinants of health between participants residing in economically disadvantaged and advantaged communities (defined by zip codes) will be compared by comparing responses to questionnaires for these two populations based on the residential zip codes. This will be conducted during Part 2 of the study.
Social Determinants of Health in Participants | Approximately 90 minutes
  Patient-specific factors will be quantified using the PRAPARE instrument, the Accountable Health Communities Health-Related Social Needs Screening Tool, and supplemental questions data collected from Part 1 of the study to compare social determinants of health among participants. This will be conducted during Part 2 of the study.
Social Determinants of Health in Participants' Communities | Approximately 90 minutes
  Community-specific factors will be quantified using the PRAPARE instrument, the Accountable Health Communities Health-Related Social Needs Screening Tool, and supplemental questions data collected from Part 1 of the study to compare social determinants of health within the participants' communities. This will be conducted during Part 2 of the study.
Comparisons of Treatment Timelines Among Low Income and High Income Communities | Approximately 90 minutes
  Time to presentation, treatment initiation, and extent of surgery for patients will be obtained from Wake Forest Baptist Comprehensive Cancer Center Registry and compared based on economically disadvantaged and advantaged communities.
Number of Low Income to High Income Community Participants | Approximately 90 minutes
  Participants will be categorized as coming from a low income community of high income community zip code through use of the CDC census data that details median household income for the zip codes provided by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Roy E. Strowd, III, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No